CLINICAL TRIAL: NCT01141608
Title: NIDA CTN Protocol 0037: Stimulant Reduction Intervention Using Dosed Exercise (STRIDE)
Brief Title: Exercise as a Treatment for Substance Use Disorders Protocol
Acronym: STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 122009-043; 5U10DA020024-05 (NIH)
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Stimulant Abuse and Dependence
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vigorous Intensity High Dose Exercise (Experimental): Usual Care Augmented with Vigorous Intensity High Dose Exercise
  Interventions: Other: Vigorous Intensity High Dose Exercise
- Health Education Intervention (Experimental): Health Education Intervention
  Interventions: Other: Health Education Intervention

INTERVENTIONS:
Other: Vigorous Intensity High Dose Exercise — Participants randomized to the exercise condition will begin with supervised exercise sessions 3 times per week during the 12-week acute phase of the study. Supervised sessions will be conducted as one-on-one (i.e., individual) sessions. Vigorous intensity high dose exercise will be prescribed at a dose of 12 kcal/kg/week (KKW), with intensity ranging from 70-85% maximal heart rate.
  Other Names: Exercise
  Arms: Vigorous Intensity High Dose Exercise
Other: Health Education Intervention — Participants randomized to the health education condition will also begin with visits 3 times per week during the 12-week acute phase. The health education sessions will be conducted as one-on-one (i.e., individual) sessions. Health education sessions will consist of information on health-related topics distributed via methods such as didactics, audio and video materials, and written materials.
  Other Names: Exercise
  Arms: Health Education Intervention

SUMMARY:
The purpose of this study is to investigate if health interventions (intensive exercise or health education) can be used to help improve substance abuse treatment. The primary objective of this protocol is to compare percent days of abstinence between Vigorous Intensity High Dose exercise (VIHD) and Health Education Intervention (HEI) groups based on stimulant (i.e., cocaine, methamphetamine, amphetamine, or other stimulant, excluding caffeine and nicotine) use during a 12-week acute phase.

DETAILED DESCRIPTION:
This study is designed as a two-group, randomized controlled trial to test the effectiveness of the addition of exercise and health education to treatment as usual in improving drug treatment outcomes in 330 eligible and interested participants who provide informed consent at 8-10 sites across the nation. These participants will be randomized to one of two treatment arms: (1) Vigorous Intensity High Dose Exercise Augmentation (VIHD): Usual Care Augmented with Vigorous Intensity High Dose Exercise or (2) Health Education Intervention Augmentation (HEI): Usual Care Augmented with Health Education. This study will include individuals diagnosed with stimulant abuse or dependence (cocaine, methamphetamine, amphetamine or other stimulant, except caffeine or nicotine) who begin treatment while in a residential setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-65.
* Admitted to residential setting and receiving substance use treatment.
* Ability to understand and willingness to provide written informed consent.
* Agree to remain in facility for authorized treatment of about 21-30 days.
* Willing to provide contact information.
* Self-reported use of stimulant drug (cocaine, methamphetamine, amphetamine, or other stimulant, excluding caffeine and nicotine) within the 30 days prior to admission for treatment.
* Meets DSM-IV criteria for substance abuse or dependence for stimulants (cocaine, methamphetamine, amphetamine, or other stimulant, excluding caffeine and nicotine) within the last 12 months.
* Medical clearance with protocol-defined stress testing (in accordance with American College of Sports Medicine (ACSM) guidelines) from protocol approved medical personnel. Details of guidelines and related testing protocol are provided in the study Manual of Procedures.
* Body mass index (BMI)≤40 kg/m2 or BMI 40 >kg/m2 and cleared by medical personnel to exercise.
* Able to comprehend and communicate in English.

Exclusion Criteria:

* Evidence of general medical condition or other abnormality that contraindicates use of exercise, based on the Medical Screening Visit.
* Current opiate dependence.
* Currently considered a high suicide risk and/or high risk for being unable to complete the study due to the need for psychiatric hospitalization, suicide attempts or suicidality, significant self-mutilation, or other self-injurious or destructive behavior based on the judgment of the site PI, medical personnel, or designee.
* Pregnancy.
* Significant physical activity, defined as aerobic exercise more than 3 times per week for 20 minutes or more, completed consistently for the three months prior to study enrollment.
* Current psychotic disorder. Other comorbid psychiatric diagnosis that, in the investigator's judgment, will pose a safety issue or make it difficult for the participant to understand or complete the intervention.
* Concomitant treatments: beta blockers; methadone, buprenorphine, or any other opioid replacement therapies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H Trivedi, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (9):
- United States (9):
  - Arapahoe House, Denver, Colorado
  - Gateway Community Services, Jacksonville, Florida
  - Gibson Recovery Center, Inc., Cape Girardeau, Missouri
  - St. Luke's-Roosevelt, New York, New York
  - Penn Presbyterian, Philadelphia, Pennsylvania
  - Charleston VAMC, Charleston, South Carolina
  - Morris Village, Columbia, South Carolina
  - Nexus Recovery, Inc., Dallas, Texas
  - Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
"Per CTN policy, study data is shared within 18-months of study completion. Data that has been shared has been completely de-identified to prevent linkages to individual research participants. This includes removal of all Personal Health Information (PHI) and indirect identifiers that are not listed as PHI but could lead to 'deductive disclosure' such as comment fields and site numbers."
Supporting Information: Study Protocol
Time Frame: 18 months following study completion.
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Derived] Jha MK, Schatzberg A, Minhajuddin A, Chin Fatt C, Mayes TL, Trivedi MH. Cross-Sectional Associations Among Symptoms of Pain, Irritability, and Depression and How These Symptoms Relate to Social Functioning and Quality of Life: Findings From the EMBARC and STRIDE Studies and the VitalSign6 Project. J Clin Psychiatry. 2021 Apr 13;82(3):20m13740. doi: 10.4088/JCP.20m13740. PMID 34000130
- [Derived] Trombello JM, Killian MO, Liao A, Sanchez K, Greer TL, Walker R, Grannemann B, Rethorst CD, Carmody T, Trivedi MH. Psychometrics of the Self-Report Concise Associated Symptoms Tracking Scale (CAST-SR): Results From the STRIDE (CTN-0037) Study. J Clin Psychiatry. 2018 Mar/Apr;79(2):17m11707. doi: 10.4088/JCP.17m11707. PMID 29325238
- [Derived] Trivedi MH, Greer TL, Rethorst CD, Carmody T, Grannemann BD, Walker R, Warden D, Shores-Wilson K, Stoutenberg M, Oden N, Silverstein M, Hodgkins C, Love L, Seamans C, Stotts A, Causey T, Szucs-Reed RP, Rinaldi P, Myrick H, Straus M, Liu D, Lindblad R, Church T, Blair SN, Nunes EV. Randomized Controlled Trial Comparing Exercise to Health Education for Stimulant Use Disorder: Results From the CTN-0037 STimulant Reduction Intervention Using Dosed Exercise (STRIDE) Study. J Clin Psychiatry. 2017 Sep/Oct;78(8):1075-1082. doi: 10.4088/JCP.15m10591. PMID 28199070
- [Derived] Warden D, Sanchez K, Greer T, Carmody T, Walker R, Dela Cruz A, Toups M, Rethorst C, Trivedi MH. Demographic and clinical characteristics of current comorbid psychiatric disorders in a randomized clinical trial for adults with stimulant use disorders. Psychiatry Res. 2016 Dec 30;246:136-141. doi: 10.1016/j.psychres.2016.09.007. Epub 2016 Sep 15. PMID 27693866
- [Derived] Trivedi MH, Greer TL, Grannemann BD, Church TS, Somoza E, Blair SN, Szapocznik J, Stoutenberg M, Rethorst C, Warden D, Ring KM, Walker R, Morris DW, Kosinski AS, Kyle T, Marcus B, Crowell B, Oden N, Nunes E. Stimulant reduction intervention using dosed exercise (STRIDE) - CTN 0037: study protocol for a randomized controlled trial. Trials. 2011 Sep 19;12:206. doi: 10.1186/1745-6215-12-206. PMID 21929768

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vigorous Intensity High Dose Exercise | Health Education Intervention
Started | 152 | 150
Completed | 152 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vigorous Intensity High Dose Exercise | Health Education Intervention | Total
Number analyzed (Participants) | 152 | 150 | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 152 | 150 | 302
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (10) | 39.5 (11) | 39 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 58 | 121
  Male | 89 | 92 | 181
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 152 | 150 | 302

OUTCOME MEASURES:

1. Primary Outcome: Percent Days Abstinent
Description: Percent days of abstinence based on stimulant (i.e., cocaine, methamphetamine, amphetamine, or other stimulant, excluding caffeine and nicotine) use during the 12-week acute phase. Days of abstinence will be measured during days 22-84, since it is anticipated that most individuals will be in a highly structured environment during the first 21 days of the study, and therefore would have little opportunity to use substances (i.e., the groups are not likely to differ during this time period). Measured by the Timeline Follow Back (TLFB) and aided by urine drug screen collected three times/week.
Time Frame: single value calculated based on TLFB data during days 22-84
Population: Mean percent stimulant abstinence days based on Timeline Follow back and Eliminate Contradiction (ELCON) algorithm adjustment.
Measure: Mean (Standard Deviation); unit: Percentage of Days
Groups:
- Vigorous Intensity High Dose Exercise: Participants randomized to Exercise completed supervised exercise sessions 3 times per week during the 12-week acute phase. Exercise was prescribed at a dose of 12 kcal/kg/week (KKW), with intensity ranging from 70-85% of maximal heart rate (HRmax).
- Health Education Intervention: Participants randomized to Health Education also completed 3 visits per week during the 12-week acute phase. Health Education consisted of one-on-one sessions in which information on health-related topics (e.g., cancer, heart disease, mental health) was distributed via didactics, websites, audio, video, and written materials.
Arm/Group | Vigorous Intensity High Dose Exercise | Health Education Intervention
Number analyzed (Participants) | 152 | 150
Percentage of Days
  Timeline Follow Back (TLFB) | 90.8 (16.4) | 91.6 (14.7)
  ELCON algorithm | 75.5 (27.4) | 77.2 (25.1)
Statistical Analysis 1: Comparison: Vigorous Intensity High Dose Exercise vs Health Education Intervention; Test type: Superiority or Other; p < 0.05, Linear mixed effects model

2. Secondary Outcome: Time to Relapse (Defined as Second Positive Urine Test [for Stimulants] and Use of Drugs Established by TLFB)
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Withdrawal Symptoms as Measured by the Stimulant Selective Severity Assessment (SSSA) and Craving as Measured by the Stimulant Craving Questionnaire-Brief (STCQ-Brief)
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Drug Use and Related Outcomes for All Substances (Categorized as Alcohol, Cannabinoids, Nicotine, Opioids, or Sedative/Hypnotic/Anxiolytics)
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Time to Dropout From Substance Abuse Treatment
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Drug Use and Related Outcomes During the Entire Course of the Study (i.e., Randomization to 9 Months)
Time Frame: 9 months
Reporting Status: Not Posted

7. Secondary Outcome: Examination of Additional Health Benefits (in Sleep, Cognitive Function, Mood, Quality of Life and Anhedonia, and Weight Gain)
Time Frame: 9 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Vigorous Intensity High Dose Exercise | Health Education Intervention
Serious Adverse Events (participants affected / at risk) | 19/152 | 21/150
Other Adverse Events (participants affected / at risk) | 79/152 | 28/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vigorous Intensity High Dose Exercise (N=152) | Health Education Intervention (N=150)
Medical condition (Surgical and medical procedures) | 19 (26) | 21 (24)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vigorous Intensity High Dose Exercise (N=152) | Health Education Intervention (N=150)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrythmia (Cardiac disorders) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
chest discomfort (General disorders) | 3 (3) | 0 (0)
chest pain (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest apin (General disorders) | 0 (0) | 1 (1)
oedema peripheral (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abcess (Infections and infestations) | 0 (0) | 1 (1)
Brochitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis cryptosporidial (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Tooth abcess (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat Stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure diastolic decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (17) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculo skeleton pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 2 (2) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1)
Post Traumatic stress Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal Behavior (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 4 (4) | 3 (3)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Victim of Crime (Social circumstances) | 1 (1) | 0 (0)
Victim of homicide (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
victim of sexual abuse (Social circumstances) | 1 (1) | 0 (0)
Sinus Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment of less severe group and differential adherence rates in the treatment arms are limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No